CLINICAL TRIAL: NCT07237373
Title: Percutaneous Thermo-ablation for the Treatment of Benign Thyroid Nodules: a Prospective Multicentric Study
Acronym: BIRRO-TA
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other); AZ Sint-Jan AV (Other)
Responsible Party: Sponsor
Other Study IDs: ONZ-2025-0427
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Benign Thyroid Nodule
Keywords: benign thyroid nodule; radiofrequency ablation; interventional radiology; percutaneous thermoablation
MeSH Terms: interventions — Catheter Ablation; Radiofrequency Ablation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Benign thyriod nodules: Subjects with symptomatic benign thyroid nodules with compressive/cosmetic complaints OR autonomously functioning thyroid nodules with subclinical hyperthyreosis or thyrotoxicosis proven on scintigraphy.
  Interventions: Device: Percutaneous radiofrequency ablation

INTERVENTIONS:
Device: Percutaneous radiofrequency ablation — RFA uses an electric field, produced by a radiofrequency generator connected to an internally cooled electrode needle, leading to frictional agitation at the ionic level and to heat generation (Joule effect). The electrode is introduced under US guidance into the target nodule, and a continuous repositioning of the applicator ("moving shot" or "multiple overlapping shot" technique). The localized heating causes necrosis and shrinkage of the thyroid nodule without damaging surrounding tissues. The appearance of hyperechoic signals close to the electrode tip indicates the development of tissue changes and air formation, while a steep rise in tissue impedance demonstrates the achievement of tissue necrosis
  Other Names: RFA; radiofrequency ablation

SUMMARY:
The goal of this observational study is to learn if radiofrequency ablation (RFA), a minimally invasive thermoablation technique, can safely reduce symptoms and improve quality of life in adults with symptomatic benign thyroid nodules or autonomously functioning thyroid nodules.

The main questions it aims to answer are:

* Does RFA improve health-related quality of life (HRQoL) as measured by the ThyPRO-39 questionnaire?
* Does RFA effectively reduce nodule volume and related symptoms (compressive or cosmetic)?

Participants will:

* Undergo a radiofrequency ablation procedure of the thyroid nodule performed under ultrasound guidance in an outpatient setting.
* Complete quality of life questionnaires (ThyPRO-39) before treatment and at follow-up visits.

Attend follow-up visits at 1, 3, 6, and 12 months with:

* Ultrasound assessments of the thyroid nodule
* Symptom and cosmetic scoring
* Blood tests to monitor thyroid function
* Safety checks for possible complications

DETAILED DESCRIPTION:
Benign thyroid nodules are highly prevalent in the adult population. While most remain asymptomatic, some patients experience compressive symptoms, cosmetic concerns, or hyperthyroidism due to autonomously functioning nodules. Standard therapy is hemithyroidectomy or total thyroidectomy, which is effective but associated with risks such as hypothyroidism, nerve injury, visible scarring, and increased health care costs. As a result, minimally invasive, nonsurgical alternatives are being actively investigated.

Radiofrequency ablation (RFA) is a percutaneous thermoablation technique performed under ultrasound guidance using a cooled electrode needle. Heat generated at the electrode tip induces localized necrosis within the target nodule, leading to progressive shrinkage while sparing surrounding thyroid tissue. In most cases, the procedure is carried out under local anesthesia in an outpatient setting, with an average duration of 15-40 minutes. The "moving shot" technique is typically employed, allowing precise ablation of large nodules in multiple overlapping steps.

International guidelines from the European Thyroid Association (ETA) and the Cardiovascular and Interventional Radiological Society of Europe (CIRSE) recommend RFA as an alternative for patients with benign thyroid nodules who present with compressive symptoms, cosmetic complaints, or autonomously functioning thyroid nodules not suitable for surgery or radioactive iodine.

This multicenter prospective observational study will investigate the clinical effectiveness and safety of RFA in routine practice. The primary outcome is health-related quality of life (HRQoL), assessed by the validated ThyPRO-39 instrument. Secondary outcomes include technical efficacy (≥50% volume reduction rate), symptom and cosmetic improvement, stability of thyroid function, and safety endpoints based on the CIRSE classification of complications.

Participants will undergo standardized baseline evaluation including ultrasound, cytology, and thyroid function testing. Follow-up visits are scheduled at 1, 3, 6, and 12 months, with systematic assessments of nodule characteristics, laboratory values, patient-reported outcomes, and complications. Technical success and regrowth will be defined according to internationally accepted thresholds.

By collecting prospective multicenter data, this study aims to generate high-quality evidence on the role of RFA in the treatment of benign thyroid nodules. The results are expected to strengthen the scientific and economic case for adopting RFA as a reimbursable, minimally invasive therapy in clinical practice, while contributing to the long-term body of literature on patient-centered outcomes in thyroid disease.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* 'Eastern Cooperative Oncology Group' (ECOG) performance status of 0 or 1
* Symptomatic benign thyroid nodules with compressive/cosmetic complaints OR autonomously functioning thyroid nodules with subclinical hyperthyreosis or thyrotoxicosis proven on scintigraphy.
* No cutoff in nodule size.
* Solid component > 20%, and benign cytology (Bethesda II) in 1 (EUTIRADS 3) or 2 (EUTIRADS 4) separate cytological assessments. In the case of a proven "hot" nodule on scintigraphy, no biopsy is required.

Exclusion Criteria:

* <18y
* Purely cystic nodule
* Severe comorbidity which limits the further life expectancy of the patient to < 2 years (opinion of the physician)
* Malignancies <2 years ago except for non-melanoma skin cancer and non-muscle invasive bladder cancer.
* Lack of compliance
* Malignant or suspicious thyroid nodules or nodules that are confluent in a compressive lobar mass
* Contralateral vocal cord paralysis
* Anticoagulant therapy that could not be suspended
* Unresolvable coagulation disorders
* Absence of consent of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants will be selected from the following Belgian hospitals: Ghent University Hospital, University Hospital Leuven, AZ Sint Jan Brugge.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2029-12-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Health related Quality Of Life (HRQoL) | From baseline (before treatment) to 12 months after the radiofrequency ablation procedure, with assessments at baseline, 1 month, 3 months, 6 months, and 12 months
  HRQoL will be assessed by the change in Thyroid-Related Patient-Reported Outcome 39 (ThyPRO-39) score from baseline to 1-year follow-up. The ThyPRO-39 is a thyroid-specific quality of life instrument covering 13 domains of QoL validated for patients with benign thyroid disease. The ThyPRO-39 includes scales assessing the following: goiter symptoms, eye symptoms, hyperthyroid symptoms, hypothyroid symptoms, tiredness, cognitive complaints, anxiety, depressivity, emotional susceptibility, impaired social life, impaired daily life, appearance, and overall QoL. Each item is rated on a Likert scale (0-4) from 0 = "no symptoms/problems" to 4 = "severe symptoms/problems." Scores are then transformed to yield 13 0-100 scales, where a higher score indicates worse health-related QoL

SECONDARY OUTCOMES:
Symptom score | From baseline (before treatment) to 12 months after the radiofrequency ablation procedure, with assessments at baseline, 1 month, 3 months, 6 months, and 12 months.
  Registered on a Visual Analog Scale (VAS), ranging from 0 to 10, where 0 indicates "no symptoms" and 10 indicates "worst imaginable symptoms".
Cosmetic score | From baseline (before treatment) to 12 months after the radiofrequency ablation procedure, with assessments at baseline, 1 month, 3 months, 6 months, and 12 months.
  Assessed during physical examination; ranging from 1 to 4, where 1 graded as no palpable mass, 2 graded as a palpable mass without cosmetic issue, 3 graded as a cosmetic problem on swallowing, and 4 as a readily detected cosmetic problem.
Number of Participants with Treatment-Related Adverse Events | From baseline (before treatment) to 12 months after the radiofrequency ablation procedure, with assessments at baseline, 1 month, 3 months, 6 months, and 12 months.
  Safety will be measured based on the presence of minor or major complications. Major and minor complications are those defined by the Society of Interventional Radiology.
Volume Reduction Rate (VRR) | From baseline (before treatment) to 12 months after the radiofrequency ablation procedure, with assessments at baseline, 1 month, 3 months, 6 months, and 12 months.
  Calculated as VRR (%) = (initial volume - final volume) ÷ initial volume × 100
Technical efficacy | From baseline (before treatment) to 12 months after the radiofrequency ablation procedure, with assessments at baseline, 1 month, 3 months, 6 months, and 12 months.
  Defined as a VRR ≥50%. Regrowth is defined as an increase in nodule volume to at least 150% of the minimum recorded volume during the follow-up period.
Thyroid function | From baseline (before treatment) to 12 months after the radiofrequency ablation procedure, with assessments at baseline, 1 month, 3 months, 6 months, and 12 months.
  Evaluation of thyroid function, including serum TSH, free T4 (FT4), and free T3 (FT3) levels

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - AZ Sint-Jan Brugge, Bruges
  - UZ Leuven, Leuven

REFERENCES:
- [Background] Shein-Chung Chow JS, Hansheng Wang, Yuliya Lokhnygina. Sample Size Calculations in Clinical Research. 3rd Edition ed2017.
- [Background] Nordqvist SF, Boesen VB, Rasmussen AK, Feldt-Rasmussen U, Hegedus L, Bonnema SJ, Cramon PK, Watt T, Groenvold M, Bjorner JB. Determining minimal important change for the thyroid-related quality of life questionnaire ThyPRO. Endocr Connect. 2021 Mar;10(3):316-324. doi: 10.1530/EC-21-0026. PMID 33617467
- [Background] Uslar V, Becker C, Weyhe D, Tabriz N. Thyroid disease-specific quality of life questionnaires - A systematic review. Endocrinol Diabetes Metab. 2022 Sep;5(5):e357. doi: 10.1002/edm2.357. Epub 2022 Jul 20. PMID 35856310
- [Background] Watt T, Bjorner JB, Groenvold M, Cramon P, Winther KH, Hegedus L, Bonnema SJ, Rasmussen AK, Ware JE Jr, Feldt-Rasmussen U. Development of a Short Version of the Thyroid-Related Patient-Reported Outcome ThyPRO. Thyroid. 2015 Oct;25(10):1069-79. doi: 10.1089/thy.2015.0209. Epub 2015 Aug 26. PMID 26214034
- [Background] Reuters KB, Mamone MCOC, Ikejiri ES, Camacho CP, Nakabashi CCD, Janovsky CCPS, Yang JH, Andreoni DM, Padovani R, Maciel RMB, Vanderlei FAB, Biscolla RPM. Bethesda Classification and Cytohistological Correlation of Thyroid Nodules in a Brazilian Thyroid Disease Center. Eur Thyroid J. 2018 Jun;7(3):133-138. doi: 10.1159/000488104. Epub 2018 Apr 27. PMID 30023345
- [Background] Filippiadis DK, Binkert C, Pellerin O, Hoffmann RT, Krajina A, Pereira PL. Cirse Quality Assurance Document and Standards for Classification of Complications: The Cirse Classification System. Cardiovasc Intervent Radiol. 2017 Aug;40(8):1141-1146. doi: 10.1007/s00270-017-1703-4. Epub 2017 Jun 5. PMID 28584945
- [Background] Russ G, Bonnema SJ, Erdogan MF, Durante C, Ngu R, Leenhardt L. European Thyroid Association Guidelines for Ultrasound Malignancy Risk Stratification of Thyroid Nodules in Adults: The EU-TIRADS. Eur Thyroid J. 2017 Sep;6(5):225-237. doi: 10.1159/000478927. Epub 2017 Aug 8. PMID 29167761
- [Background] Wang JF, Wu T, Hu KP, Xu W, Zheng BW, Tong G, Yao ZC, Liu B, Ren J. Complications Following Radiofrequency Ablation of Benign Thyroid Nodules: A Systematic Review. Chin Med J (Engl). 2017 Jun 5;130(11):1361-1370. doi: 10.4103/0366-6999.206347. PMID 28524837
- [Background] Hegedus L, Frasoldati A, Negro R, Papini E. European Thyroid Association Survey on Use of Minimally Invasive Techniques for Thyroid Nodules. Eur Thyroid J. 2020 Jul;9(4):194-204. doi: 10.1159/000506513. Epub 2020 Mar 27. PMID 32903971
- [Background] Bernardi S, Dobrinja C, Fabris B, Bazzocchi G, Sabato N, Ulcigrai V, Giacca M, Barro E, De Manzini N, Stacul F. Radiofrequency ablation compared to surgery for the treatment of benign thyroid nodules. Int J Endocrinol. 2014;2014:934595. doi: 10.1155/2014/934595. Epub 2014 Jun 22. PMID 25045352
- [Background] Deandrea M, Trimboli P, Garino F, Mormile A, Magliona G, Ramunni MJ, Giovanella L, Limone PP. Long-Term Efficacy of a Single Session of RFA for Benign Thyroid Nodules: A Longitudinal 5-Year Observational Study. J Clin Endocrinol Metab. 2019 Sep 1;104(9):3751-3756. doi: 10.1210/jc.2018-02808. PMID 30860579
- [Background] Baek JH, Lee JH, Sung JY, Bae JI, Kim KT, Sim J, Baek SM, Kim YS, Shin JH, Park JS, Kim DW, Kim JH, Kim EK, Jung SL, Na DG; Korean Society of Thyroid Radiology. Complications encountered in the treatment of benign thyroid nodules with US-guided radiofrequency ablation: a multicenter study. Radiology. 2012 Jan;262(1):335-42. doi: 10.1148/radiol.11110416. Epub 2011 Oct 13. PMID 21998044
- [Background] Jeong WK, Baek JH, Rhim H, Kim YS, Kwak MS, Jeong HJ, Lee D. Radiofrequency ablation of benign thyroid nodules: safety and imaging follow-up in 236 patients. Eur Radiol. 2008 Jun;18(6):1244-50. doi: 10.1007/s00330-008-0880-6. Epub 2008 Feb 20. PMID 18286289
- [Background] Deandrea M, Sung JY, Limone P, Mormile A, Garino F, Ragazzoni F, Kim KS, Lee D, Baek JH. Efficacy and Safety of Radiofrequency Ablation Versus Observation for Nonfunctioning Benign Thyroid Nodules: A Randomized Controlled International Collaborative Trial. Thyroid. 2015 Aug;25(8):890-6. doi: 10.1089/thy.2015.0133. Epub 2015 Jul 13. PMID 26061686
- [Background] Baek JH, Lee JH, Valcavi R, Pacella CM, Rhim H, Na DG. Thermal ablation for benign thyroid nodules: radiofrequency and laser. Korean J Radiol. 2011 Sep-Oct;12(5):525-40. doi: 10.3348/kjr.2011.12.5.525. Epub 2011 Aug 24. PMID 21927553
- [Background] Baek JH, Kim YS, Lee D, Huh JY, Lee JH. Benign predominantly solid thyroid nodules: prospective study of efficacy of sonographically guided radiofrequency ablation versus control condition. AJR Am J Roentgenol. 2010 Apr;194(4):1137-42. doi: 10.2214/AJR.09.3372. PMID 20308523
- [Background] Kohlhase KD, Korkusuz Y, Groner D, Erbelding C, Happel C, Luboldt W, Grunwald F. Bipolar radiofrequency ablation of benign thyroid nodules using a multiple overlapping shot technique in a 3-month follow-up. Int J Hyperthermia. 2016 Aug;32(5):511-6. doi: 10.3109/02656736.2016.1149234. Epub 2016 Apr 28. PMID 27126512
- [Background] Park HS, Baek JH, Park AW, Chung SR, Choi YJ, Lee JH. Thyroid Radiofrequency Ablation: Updates on Innovative Devices and Techniques. Korean J Radiol. 2017 Jul-Aug;18(4):615-623. doi: 10.3348/kjr.2017.18.4.615. Epub 2017 May 19. PMID 28670156
- [Background] Kim JH, Baek JH, Lim HK, Ahn HS, Baek SM, Choi YJ, Choi YJ, Chung SR, Ha EJ, Hahn SY, Jung SL, Kim DS, Kim SJ, Kim YK, Lee CY, Lee JH, Lee KH, Lee YH, Park JS, Park H, Shin JH, Suh CH, Sung JY, Sim JS, Youn I, Choi M, Na DG; Guideline Committee for the Korean Society of Thyroid Radiology (KSThR) and Korean Society of Radiology. 2017 Thyroid Radiofrequency Ablation Guideline: Korean Society of Thyroid Radiology. Korean J Radiol. 2018 Jul-Aug;19(4):632-655. doi: 10.3348/kjr.2018.19.4.632. Epub 2018 Jun 14. PMID 29962870
- [Background] Gharib H, Hegedus L, Pacella CM, Baek JH, Papini E. Clinical review: Nonsurgical, image-guided, minimally invasive therapy for thyroid nodules. J Clin Endocrinol Metab. 2013 Oct;98(10):3949-57. doi: 10.1210/jc.2013-1806. Epub 2013 Aug 16. PMID 23956350
- [Background] Navin PJ, Thompson SM, Kurup AN, Lee RA, Callstrom MR, Castro MR, Stan MN, Welch BT, Schmitz JJ. Radiofrequency Ablation of Benign and Malignant Thyroid Nodules. Radiographics. 2022 Oct;42(6):1812-1828. doi: 10.1148/rg.220021. PMID 36190855
- [Background] Collins RA, McManus C, Kuo EJ, Liou R, Lee JA, Kuo JH. Improvement in thyroid-specific quality of life following radiofrequency ablation of benign thyroid nodules: A USA study. Surgery. 2025 Jan;177:108823. doi: 10.1016/j.surg.2024.06.063. Epub 2024 Oct 9. PMID 39384472
- [Background] Loncar I, van Dijk SPJ, van Velsen EFS, Buijk SE, Niemeijer ND, Veeken CJ, von Meyenfeldt EM, Dinkelaar W, Franssen GJH, Peeters RP, Massolt ET, Moelker A, van Ginhoven TM. Radiofrequency Ablation for Benign Symptomatic Thyroid Nodules in the Netherlands: Successful Introduction of a Minimally Invasive Treatment Option Improving Quality of Life. J Vasc Interv Radiol. 2022 May;33(5):530-537.e1. doi: 10.1016/j.jvir.2022.01.012. Epub 2022 Feb 2. PMID 35121096
- [Background] Papini E, Monpeyssen H, Frasoldati A, Hegedus L. 2020 European Thyroid Association Clinical Practice Guideline for the Use of Image-Guided Ablation in Benign Thyroid Nodules. Eur Thyroid J. 2020 Jul;9(4):172-185. doi: 10.1159/000508484. Epub 2020 Jun 8. PMID 32903999